CLINICAL TRIAL: NCT04682314
Title: B-Cell Reconstitution After Hematopoietic Stem Cell Transplantation
Acronym: B-REC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201015
Record Dates: First submitted 2020-12-07; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is a potentially curative treatment for a variety of hematological malignancies. However, patients who have received this treatment have a persistent deficit in humoral immunity up to one year post-transplant. To date, the design of new therapeutic strategies to improve immune recovery in allo-HSCT patients is still hampered by the fact that post-transplant regenerative hematopoiesis has never been studied, and more generally by our currently limited knowledge on the development and function of human B lymphocytes. The main objective of our study is to study early B-cell progenitor reconstitution after allogeneic hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* 18 years of age and older
* with hematological malignancies and subject to allogeneic HSCT
* with health insurance coverage (bénéficiaire ou ayant droit)
* having signed a written informed consent.

Inclusion criteria of donor

* 18 years of age and older
* with health insurance coverage (bénéficiaire ou ayant droit)
* having signed a specific written informed consent.

Exclusion criteria of recipient and donor

* Absence of written informed consent
* Patient or donor on AME
* Patient or donor on AME or under protection by law, tutorship or curatorship
* Pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older with hematological malignancies and subject to allogeneic HSCT
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
B cells reconstitution | at day 100 days post-transplant
  B cell clusters as assess by CyTOF technology

SECONDARY OUTCOMES:
B cells reconstitution | at 6 months post-transplant
  B cell clusters as assess by CyTOF technology
Perturbations in growth or differentiation of progenitor/precursor of B cells | at 100 days post transplant
  Perturbations in growth or differentiation of progenitor/precursor of B cells will be assessed by cytometry technology
Perturbations in growth or differentiation of progenitor/precursor of B cells | at 6 months post-transplant
  Perturbations in growth or differentiation of progenitor/precursor of B cells will be assessed by cytometry technology

IPD SHARING:
Plan to Share IPD: Undecided